CLINICAL TRIAL: NCT04670705
Title: The Prevalence of Acute Pancreatitis Episodes Among Patients With Chronic Pancreatitis and the Associated Factors
Brief Title: Relationship of CP and AP
Status: Completed | Type: Observational
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhuan Liao, Principal Investigator, Changhai Hospital
Other Study IDs: AP&CP
Record Dates: First submitted 2020-12-11; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Chronic Pancreatitis; Acute Pancreatitis
MeSH Terms: conditions — Pancreatitis, Chronic; Pancreatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: patients' characteristics — There was no intervention.

SUMMARY:
The present study aimed to determine the prevalence of AP attacks before the diagnosis of CP and further identified the potential associated factors for AP episodes.

ELIGIBILITY:
Inclusion Criteria:

* Consequent patients with a diagnosis of CP between January 2010 to December 2015
* informed consents provided

Exclusion Criteria:

* autoimmune pancreatitis (AIP)
* pancreatic cancer diagnosed within 2 years after the diagnosis of CP

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consequent patients with a diagnosis of CP were enrolled between January 2010 to December 2015 after informed consents obtained.The diagnosis of CP was established based on the findings of computed tomography, magnetic resonance imaging, or endoscopic ultrasound, in accordance with the Asia-Pacific consensus.
Sampling Method: Non-Probability Sample
Enrollment: 1022 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2020-10 (Actual)

PRIMARY OUTCOMES:
the occurrence of acute pancreatitis | Baseline (before the diagnosis of CP)
  the presence and frequency of acute pancreatitis before diagnosis of CP

IPD SHARING:
Plan to Share IPD: Undecided